CLINICAL TRIAL: NCT05569551
Title: Umbilical Cord Care in Term Neonates: The Revolutionized Role of Wondaleaf Adhesive Pouch (WLAP) in the Prevention of Neonatal Sepsis
Brief Title: Umbilical Cord Care in Term Neonates: The Role of Wondaleaf Adhesive Pouch (WLAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AIMST University Malaysia (Other)
Collaborators: Putra Medical Centre, Malaysia (Unknown); Twin Catalyst Sdn Bhd, Malaysia (Unknown)
Responsible Party: Principal Investigator, Yu Chye Wah, Professor, AIMST University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AURRB/IND/TWIN/2020/01
Record Dates: First submitted 2022-09-25; First posted 2022-10-06 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Umbilical Cord Infection; Umbilical Sepsis; Neonatal Sepsis
Keywords: Umbilical cord care; Omphalitis; Neonatal sepsis; Barrier dressing
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking on participants and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesive pouch (Experimental): Experimental group will be applied with Wondaleaf adhesive pouch to cover up the umbilical stump
  Interventions: Device: Adhesive pouch
- Conventional care (No Intervention): Control group will not be applied with Wondaleaf adhesive pouch, but the umbilical stump is managed with conventional care, by cleaning with antiseptic.

INTERVENTIONS:
Device: Adhesive pouch — Is a barrier dressing categorized under class C medical device. It is used to seal up the umbilical stump to prevent contamination until its cord detachment. It has an adhesive film that sticks to skin with a centrally located non-adhesive pouch ensuring that zero pressure is applied on the umbilicus. It is made of polyurethane, the same material as transparent intravenous cannula dressings making it hypoallergenic waterproof and breathable.
  Other Names: Wondaleaf adhesive pouch (WLAP)
  Arms: Adhesive pouch

SUMMARY:
The purpose of this study is to evaluate the efficacy of Wondaleaf Adhesive Pouch (WLAP) in the prevention of umbilical cord infection among full-term neonates.

Methods: This is a prospective double-blinded randomized controlled trial on 218 term neonates in which 109 each was randomly assigned to interventional and conventional group. The Wondaleaf Adhesive Pouch (WLAP) dressings were applied to umbilical stumps of the term neonates in interventional group by trained midwife on the first day immediate after delivery. Mothers or caregivers were taught to observe the umbilical stump the subsequent days till the stump detached. The observations are supported by photographic images taken by caregiver and evaluated by the trial team and reporting inflammation with immediately removal of WLAP or otherwise no sign of infection till the detachment of stump.

DETAILED DESCRIPTION:
Background: Neonatal death was the serious global burden with three-quarter of it was attributable to neonatal sepsis. It was estimated that the annual incidence cases have reached 1.3 million and posed significant economic impact to many low-income and middle-income countries. The purpose of this study is to evaluate the efficacy of Wondaleaf Adhesive Pouch (WLAP) in the prevention of umbilical cord infection among full-term neonates.

Methods: This is a prospective double-blinded randomized controlled trial conducted in one hospital located in state of Kedah, Malaysia on 218 term neonates in which 109 each was randomly assigned to interventional and conventional group. The Wondaleaf Adhesive Pouch (WLAP) dressings were applied to umbilical stumps of the term neonates in interventional group by trained midwife on the first day immediate after delivery. Mothers or caregivers will be taught to observe the umbilical stump the subsequent days till the stump detached. The observations are supported by photographic images taken by caregiver to be evaluated by the trial team and reporting inflammation with immediately removal of WLAP or otherwise no sign of infection till the detachment of stump.

Results and conclusion will be reported after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Normal term neonates
* Born in the study site (hospital)

Exclusion Criteria:

* Congenital abnormalities
* Apgar score less than 7
* Neonatal conditions

Ages: 1 Hour to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
Umbilical cord infection rate | From the date of randomization until the date of cord infection occurred, assessed up to 3 weeks
  Number of neonates with umbilical cord infection. Comparing the umbilical cord infection rate between experimental group and control group. If the experimental group with WLAP applied has a lower rate of infection against the published literature, then WLAP can be shown to be effective.

SECONDARY OUTCOMES:
Duration of cord detachment | From date of randomization until the date of cord detached, assessed up to 2 weeks
  Number of days for umbilical cord detachment. If the duration of cord detachment for experimental group is equal to control group, then Wondaleaf Adhesive Pouch (WLAP) has no effect on the detachment mechanism of the umbilical stump

CONTACTS AND LOCATIONS:
Overall Officials: Chye Wah Yu, PhD, Principal Investigator — AIMST University Malaysia
Locations (1):
- AIMST University Malaysia, Bedong, Kedah, Malaysia

IPD SHARING:
Plan to Share IPD: No
Not intent to share as sponsor and stakeholders involved have to agree with this plan.

REFERENCES:
- [Result] Coffey PS, Brown SC. Umbilical cord-care practices in low- and middle-income countries: a systematic review. BMC Pregnancy Childbirth. 2017 Feb 20;17(1):68. doi: 10.1186/s12884-017-1250-7. PMID 28219420
- [Result] Stewart D, Benitz W; COMMITTEE ON FETUS AND NEWBORN. Umbilical Cord Care in the Newborn Infant. Pediatrics. 2016 Sep;138(3):e20162149. doi: 10.1542/peds.2016-2149. PMID 27573092
- [Result] Leante Castellanos JL, Perez Munuzuri A, Ruiz Campillo CW, Sanz Lopez E, Benavente Fernandez I, Sanchez Redondo MD, Rite Gracia S, Sanchez Luna M. [Recommendations for the care of the umbilical cord in the newborn]. An Pediatr (Engl Ed). 2019 Jun;90(6):401.e1-401.e5. doi: 10.1016/j.anpedi.2019.01.019. Epub 2019 Apr 7. Spanish. PMID 30971383

DOCUMENTS (1):
  • Informed Consent Form (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05569551/ICF_000.pdf